CLINICAL TRIAL: NCT05540652
Title: Developing and Testing Internet-Based Mindfulness Intervention to Reduce Minority Stress and Promote HIV-Related Behavioral Health Among Young Adult Sexual Minority Men: An Open Pilot
Brief Title: Developing an Online Mindfulness-based Intervention to Reduce Minority Stress and HIV Risk Among Young Adult MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2004002698; K23AT011173 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-05

CONDITIONS: HIV; Minority Stress; Mental Health Wellness 1
Keywords: Mindfulness-based intervention; Sexual minority; LGBTQ; HIV prevention

STUDY DESIGN:
Intervention Model Description: This is a single arm trial testing an internet delivered mindfulness-based intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Based Queer Resilience (MBQR) (Experimental): This is a single arm trial testing an internet delivered mindfulness-based intervention. All enrolled participants will receive the study intervention.
  Interventions: Behavioral: Mindfulness-Based Queer Resilience (MBQR)

INTERVENTIONS:
Behavioral: Mindfulness-Based Queer Resilience (MBQR) — "Mindfulness-based Queer Resilience (MBQR)" is an internet delivered group-based, LGBTQ affirmative mindfulness program designed to address minority stress and promote mental and sexual health among young adult gay, bisexual, and queer men. The intervention group will meet once a week for up to 2.5 hours for nine weeks. Participants will receive free training in meditation, mindful movements, and in directing mindfulness-based skills towards enhancing things like stress recovery, sleep, resilience, cognitive performance and social relationships. MBQR was adapted from the Mindfulness-Based Stress Reduction program. Customization of the curriculum was developed by queer researchers and teachers, with input from the LGBTQ community.

SUMMARY:
The overall aim of the research study is to develop and test a mindfulness-based program for young adult gay, bisexual, and queer men at risk for HIV (Brown University IRB approved protocol #2004002698). Researchers have completed Aim 1 of the broader study, which was to use qualitative, community engaged methods, along with a quantitative online survey, to inform intervention development with the study population. The next phase of the intervention development (Aim 2 - registered here), involves seeking feedback on the developed mindfulness program through an open-pilot with 18 participants from the same study population (young adult gay, bisexual, and queer men at risk for HIV).

DETAILED DESCRIPTION:
In 2017, gay, bisexual, and other men who have sex with men (MSM) made up 70% of new HIV infections in the U.S., and young adult MSM (age 18-34; YMSM) account for the majority of HIV cases. YMSM also experience prevalent, often co-occurring mental health issues, including depression, anxiety, and substance use, creating a "syndemic" condition surrounding HIV risk and suboptimal HIV testing.

A key driver of such disparities experienced by YMSM is minority stress. Experiences of identity-based discrimination lead to internalized stigma and maladaptive coping (e.g., emotion dysregulation, avoidant coping, impulsivity) The "downstream" effects of minority stress are poor mental health (depression and anxiety), increased sexual risk, and lack of engagement in key health services such as HIV testing due to anxiety related to identity disclosure to providers and anticipation of stigmatizing encounters. Recent evidence also suggests discrimination exposure is linked to heightened physiological stress response (cortisol level) that represents depletion of coping resources and increased risk for development of stress-linked psychological disorders (depression, anxiety). Therefore, reducing minority stress represents a promising transdiagnostic approach to reduce the burden of HIV and mental health issues experienced by YMSM.

Research suggests that Mindfulness-Based Interventions (MBIs) target mechanisms relevant to minority stress, including self-acceptance, emotional dysregulation, and avoidant coping. Therefore, as an individual-level intervention, MBIs may serve as an innovative HIV prevention intervention by lowering the syndemic risk among YMSM through reducing psychological symptoms, improving coping, and enhancing HIV-related behavioral health. However, no evidence-based MBIs have been tested for HIV prevention, and clinical and research evidence suggests further adaptation is warranted to improve its relevance and optimize engagement for YMSM.

This study aims to develop an internet-delivered MBI to address minority stress and its negative HIV-related health consequences experienced by YMSM. Specifically, the researchers propose to adapt, refine, and pilot-test an evidence-based MBI, Mindfulness-based Stress Reduction (MBSR), to promote mental and sexual health and HIV testing engagement among distressed, high-risk YMSM. Aims 1-3 will support the subsequent production and evaluation of the adapted intervention. To maximize reach, scalability, and availability to a population that experience challenges seeking in-person counseling and health services, the intervention will also be adapted for internet-based delivery.

Aim 1. (Previously Completed) Adapt MBSR for distressed, high-risk YMSM using internet delivery, guided by the ADAPT-ITT model. Researchers conducted iterative phases of formative research including online-based focus groups with YMSM, solicitation of feedback from stakeholders, and revision of intervention protocols. This process resulted in the first-draft of an internet-delivered, mindfulness-based intervention protocol for use with YMSM, known as "Mindfulness-Based Queer Resilience (MBQR)".

Aim 2. (This is the focus of this Clinical Trial Registration) Refine intervention protocol by administering adapted materials to distressed, high-risk YMSM (n=18) through internet-based open pilot and gather feedback. Following integration of feedback, this process will result in a finalized protocol of an internet-delivered, mindfulness-based intervention protocol for YMSM.

Aim 3. (Future research) Examine the feasibility and acceptability of an internet-delivered mindfulness-based intervention (iMBI) for HIV prevention. A sample of 40 distressed, high-risk YMSM will be randomized into the adapted iMBI or an active control condition. Primary outcome will be intervention feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male at birth
* Being 18 to 34 years of age
* Identify as a cisgender man
* Reside in the United States
* Can read and speak in English
* Engaged in condomless anal sex with another man in the past 6-months
* Endorse distress, measured by the PHQ-9 and GAD-7
* Possess a device (phone, tablet, computer) that allows for online conferencing
* HIV-negative or status unknown (self-report)

Exclusion Criteria: Participants will be excluded from the study if they are determined to have symptoms preventing them from giving meaningful consent or study activities such as:

* Significant cognitive impairment
* Psychosis
* Imminent suicidal risk
* Substance abuse

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shufang Sun, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Following data collection, cleaning, and analysis, we plan to publish de-identified quantitative data at an open science data repository (e.g., Open Science Framework). De-identified qualitative data will be available upon request to the study PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Fall 2023

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-Based Queer Resilience (MBQR)
Started | 19
Completed | 18 (1 participant was lost to follow-up between intervention initiation and post-intervention assessment)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mindfulness-Based Queer Resilience (MBQR)
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (4.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12
  Nonbinary, gender non-conforming, genderqueer, genderfluid | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 1
  Race: Asian | 3
  Race: Black | 1
  Race: Native Hawaiian and other Pacific Islander | 0
  Race: White | 11
  Race: Other | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Sexual Orientation [Count of Participants; unit: Participants]
  Bisexual | 0
  Gay | 16
  Pansexual | 1
  Straight | 0
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Online Mindfulness-Based Queer Resilience as Measured by Recruitment Rates
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Feasibility will be assessed via three measures. One measure of feasibility will be participant recruitment rates. See other primary outcomes for other measures used.
Time Frame: Baseline
Population: Overall Number of Participants Analyzed represents number of participants eligible for study from the online screener.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Queer Resilience (MBQR)
Number analyzed (Participants) | 71
Participants | 19

2. Primary Outcome: Feasibility of Online Mindfulness-Based Queer Resilience as Measured by Retention Rates
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Feasibility will be assessed via three measures. One measure of feasibility will be participant retention rates (i.e., as measured by attrition). See other primary outcomes for other measures used.
Time Frame: Through study completion, an average of 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Queer Resilience (MBQR)
Number analyzed (Participants) | 19
Participants
  Post-intervention follow-up | 18
  Exit interview | 15

3. Primary Outcome: Feasibility of Online Mindfulness-Based Queer Resilience as Measured by Session Attendance and Home Practice Completion
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. Feasibility was assessed via three measures. One measure of feasibility is engagement with the intervention content, which is calculated using the average number of weeks that participants (1) attended the MBQR sessions and (2) completed the home practices, reported here.
Time Frame: Through intervention completion, an average of 2 months
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Mindfulness-Based Queer Resilience (MBQR)
Number analyzed (Participants) | 19
Weeks
  Enactment of treatment skills | 5.84 (2.14)
  Session Attendance | 5.32 (2.29)

4. Primary Outcome: Acceptability of Online Mindfulness-Based Queer Resilience as Measured by the Client Satisfaction Questionnaire
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. One measure of acceptability will be via acceptability ratings using the validated 8-item Client Satisfaction Questionnaire (CSQ-8). Scores for the CSQ-8 range from 8 to 32, with higher values indicating higher satisfaction. See other primary outcomes for other measures used.
Time Frame: Post-intervention assessment (i.e., at 8 weeks, after intervention delivery)
Population: 1 participant was lost to follow-up before the post-intervention follow-up.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mindfulness-Based Queer Resilience (MBQR)
Number analyzed (Participants) | 18
Scores on a scale | 26.17 (5.17)

5. Primary Outcome: Acceptability of Online Mindfulness-Based Queer Resilience as Measured by a Session Evaluation Form
Description: The primary aim of the study is to evaluate feasibility and acceptability of Mindfulness-Based Queer Resilience. One measure of acceptability will be via acceptability ratings using the session evaluation form. The survey includes 6 open-ended questions and 10 items on a 4-point Likert scale ranging from 1 (strongly agree) to 4 (strongly disagree). Example Likert items include "The MBQR program was well organized". Scores for the session evaluation form range from 10 to 40, with lower values indicating higher satisfaction. See other primary outcomes for other measures used.
Time Frame: Post-intervention assessment (i.e., at 8 weeks, after intervention delivery)
Population: 1 participant was lost to follow-up before the post-intervention follow-up.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mindfulness-Based Queer Resilience (MBQR)
Number analyzed (Participants) | 18
Scores on a scale | 16.17 (5.25)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 2 months
Arm/Group | Mindfulness-Based Queer Resilience (MBQR)
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT05540652/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT05540652/SAP_001.pdf
  • Informed Consent Form (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT05540652/ICF_002.pdf